CLINICAL TRIAL: NCT04470297
Title: Adjuvant Therapeutic Effects of Melatonin Agonist on Hospitalized Patients With Confirmed or Suspected COVID-19
Brief Title: Melatonin Agonist on Hospitalized Patients With Confirmed or Suspected COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Principal Investigator, Ronaldo Delmonte Piovezan, PhD, Associação Fundo de Incentivo à Pesquisa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MELCOV2020
Record Dates: First submitted 2020-07-12; First posted 2020-07-14 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Covid19; Lung Injury
Keywords: COVID-19; Acute Distress Respiratory Syndrome; Melatonin
MeSH Terms: conditions — COVID-19; Lung Injury; Respiratory Distress Syndrome | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): A placebo with the same physical characteristics of the experimental drug pill will be administered at the same time and daily schedule as the experimental intervention for 10 days.
  Interventions: Drug: Ramelteon 8mg
- Ramelteon (Experimental): A pill containing ramelteon 8mg will be administered daily at bedtime for 10 days.
  Interventions: Drug: Ramelteon 8mg

INTERVENTIONS:
Drug: Ramelteon 8mg — Standard care combined with oral placebo or ramelteon 8mg at bedtime for 10 days

SUMMARY:
COVID-19 is impacting on health systems in Brazil and worldwide. Reducing the risk of clinical deterioration and prolonged disease duration in hospitalized patients with COVID-19 may alleviate the burden caused by the pandemic. Melatonin (N-acetyl-5-methoxytryptamine) has demonstrated antiapoptotic, antioxidative, and anti-inflammatory roles and has been suggested as a potential protector against organ injuries and even mediate lower mortality rates after polymicrobial sepsis in animal models. Melatonin agonists may modulate protective effects against acute lung injury and play a clinical role in individuals with SARS-CoV-2 infection. The investigators proposed a clinical trial testing the effects of ramelteon 8mg in hospitalized patients with COVID-19.

DETAILED DESCRIPTION:
The severe acute respiratory syndrome coronavirus 2 (SARS CoV-2) pandemic, also denominated Coronavirus Disease 2019 (COVID-19), is currently challenging health systems in Brazil and worldwide. The mortality rate of confirmed cases of COVID-19 in Brazil seems to be close to twice that of countries like Germany and Canada. (1-3) The resulted viral interstitial pneumonia can lead to severe hypoxemic respiratory failure, overcrowded intensive care units (ICUs), shortages of equipment and personnel, and increased mortality. (4-6)

Some reasons for higher mortality risk in Brazil can be related to an increased propensity of clinical worsening in hospitalized patients. Consequently, reducing the risk of clinical deterioration and prolonged disease duration in hospitalized patients with mild-to-moderate COVID-19 has become a priority to reduce the burden of such pandemic and the admission to ICUs. However, to our knowledge, few and complex specific interventions have been tested targeting outcomes related to a reduction of the immediate risk of severe disease and prolonged hospitalization in inpatients with mild-to-moderate clinical signs and symptoms.

Melatonin (N-acetyl-5-methoxytryptamine) is a hormone synthesized mainly by the pineal gland and also by other nonendocrine organs, including the immune system. Among its multiple properties, melatonin has demonstrated antiapoptotic, antioxidative, and anti-inflammatory roles exerted via both receptor-dependent and receptor-independent signalling cascades. (7,8) It has been suggested that melatonin receptors activation protects against organ injuries. (9-10). Additionally, melatonin receptors can mediate lower mortality rates after polymicrobial sepsis in animal models. (11)

Melatonin potentially modulates immune response by enhancing the secretion of anti-inflammatory cytokines including IL-10, which is involved in the Th2-like immune response. (12) IL-10 has effects on a myriad of cell types and, in lung cells under damaging circumstances, its production turns undermined. (13) Recent findings indicated that melatonin receptors are modulators of protective effects against acute lung injury induced by the ventilator in rats through the up-regulation of IL-10 production. (14) This evidence upsurged testing the effects of ramelteon, a potent and highly selective agonist of high-affinity melatonin receptors 1 (MT1) and MT2, which further displays antioxidative and anti-inflammatory properties. (15-17) Melatonin agonism may play a clinical role in individuals with acute lung injuries, including those induced by SARS-CoV-2 infection, which has not yet been investigated. The investigators designed a clinical trial testing standard care versus ramelteon 8mg under diverse clinical and laboratory outcomes related to the COVID-19 in hospitalized patients with this condition.

References

1. Robert Koch Institut. Coronavirus Disease 2019 (COVID-19) Daily Situation Report of the Robert Koch Institute. Available from: https://www.rki.de/DE/Content/InfAZ/N/Neuartiges_Coronavirus/Situationsberichte/Gesamt.html Updated 14.05.20
2. DATASUS. Ministério da Saúde do Brasil. Available from: https://covid.saude.gov.br/. Atualizada em: 14/05/2020
3. Government of Canada. Coronavirus Disease 2019 (COVID-19): Daily Epidemiology Update. Available from: https://www.canada.ca/en/public-health/services/diseases/2019-novel-coronavirus-infection.html?topic=tilelink#a1. Updated 14.05.20.
4. P.H.S. Pelicioni, S.R. Lord. COVID-19 will severely impact older people's lives, and in many more ways than you think!. Braz J Phys Ther, (2020), http://dx.doi.org/10.1016/j.bjpt.2020.04.005
5. [3] R.D. Branson, D.R. Hess, L. Rubinson. SARS CoV-2: Guidance Document. American Association for Respiratory Care, (2020),
6. World Health Organization. Coronavirus Disease 2019 (COVID-19) Situation Report 46. (2020)
7. Jockers R, Delagrange P, Dubocovich ML, Markus RP, Renault N, Tosini G, Cecon E, Zlotos DP. Update on melatonin receptors: IUPHAR Review 20. Br J Pharmacol. 2016;173:2702-2725. doi: 10.1111/bph.13536.
8. Radogna F, Paternoster L, Albertini MC, Cerella C, Accorsi A, Bucchini A, Spadoni G, Diamantini G, Tarzia G, De Nicola M, et al. Melatonin antagonizes apoptosis via receptor interaction in U937 monocytic cells. J Pineal Res. 2007;43:154-162. doi: 10.1111/j.1600-079X.2007.00455.x.
9. Lochner A, Genade S, Davids A, Ytrehus K, Moolman JA. Short- and long-term effects of melatonin on myocardial post-ischemic recovery. J Pineal Res. 2006;40:56-63. doi: 10.1111/j.1600-079X.2005.00280.x.
10. Rezzani R, Rodella LF, Bonomini F, Tengattini S, Bianchi R, Reiter RJ. Beneficial effects of melatonin in protecting against cyclosporine A-induced cardiotoxicity are receptor-mediated. J Pineal Res. 2006;41:288-295. doi: 10.1111/j.1600-079X.2006.00368.x.
11. Fink T, Glas M, Wolf A, Kleber A, Reus E, Wolff M, Kiefer D, Wolf B, Rensing H, Volk T, Mathes AM. Melatonin receptors mediate improvements of survival in a model of polymicrobial sepsis. Crit Care Med. 2014;42:e22-e31. doi: 10.1097/CCM.0b013e3182a63e2b.
12. Ren Wenkai, Liu Gang, Chen Shuai, Yin Jie, Wang Jing, Tan Bie, Wu Guoyao, Bazer Fuller W., Peng Yuanyi, Li Tiejun, Reiter Russel J., Yin Yulong. Melatonin signalling in T cells: Functions and applications. Journal of Pineal Research. 2017;62(3):e12394. doi: 10.1111/jpi.12394.
13. Hokenson MA, Wang Y, Hawwa RL, Huang Z, Sharma S, Sanchez-Esteban J. Reduced IL-10 production in fetal type II epithelial cells exposed to mechanical stretch is mediated via activation of IL-6-SOCS3 signalling pathway. PLoS One. 2013;8:e59598. doi: 10.1371/journal.pone.0059598.
14. Wu GC, Peng CK, Liao WI, Pao HP, Huang KL, Chu SJ. Melatonin receptor agonist protects against acute lung injury induced by ventilator through up-regulation of IL-10 production. Respir Res. 2020 Mar 6;21(1):65. doi: 10.1186/s12931-020-1325-2.
15. Mathes AM, Kubulus D, Waibel L, Weiler J, Heymann P, Wolf B, Rensing H. Selective activation of melatonin receptors with ramelteon improves liver function and hepatic perfusion after hemorrhagic shock in the rat. Crit Care Med. 2008;36:2863-2870. doi: 10.1097/CCM.0b013e318187b863.
16. Shimizu N, Nozawa M, Sugimoto K, Yamamoto Y, Minami T, Hayashi T, Yoshimura K, Ishii T, Uemura H. Therapeutic efficacy and anti-inflammatory effect of ramelteon in patients with insomnia associated with lower urinary tract symptoms. Res Rep Urol. 2013;5:113-119.
17. Zhou W, Zhang X, Zhu CL, He ZY, Liang JP, Song ZC. Melatonin receptor agonists as the "Perioceutics" agents for the periodontal disease through modulation of Porphyromonas gingivalis virulence and inflammatory response. PLoS One. 2016;11:e0166442. doi: 10.1371/journal.pone.0166442

ELIGIBILITY:
Inclusion Criteria:

1. Individuals (or legally authorized representative) providing written informed consent prior to initiation of any study procedures.
2. Male or non-pregnant female adult ≥18 years of age at time of enrollment
3. Subject consents to randomization within 48 hours of hospital admission
4. Symptom duration of 14 days or less upon recruitment
5. At least one of the following:

   1. Radiographic infiltrates by imaging (chest x-ray or CT scan), OR
   2. Clinical assessment (evidence of rales/crackles on the exam) AND SpO2 ≤ 94% on room air

Exclusion Criteria:

1. Mild COVID-19 disease (minor clinical symptoms, imaging does not show signs of lung inflammation)
2. Recent history of or any in-hospital exposure to investigational medications targeting COVID-19
3. ALT/AST > 5 times the upper limit of normal.
4. Known hypersensitivity to ramelteon
5. Pregnancy
6. Severe hepatic insufficiency
7. Fluvoxamine use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Time to resolution of symptoms [National Early Warning Score 2 (NEWS2) of 0] | enrollment is day 0
  Defined as a National Early Warning Score 2 (NEWS2) of 0 maintained for 24 hours [Time Frame: Assessed daily (enrollment is day 0)] The NEWS consists of a simple aggregate scoring system based on physiological measurements, regularly registered in inpatient settings, including six parameters: respiration rate, oxygen saturation, systolic blood pressure, pulse rate, level of consciousness or new confusion, and temperature.

SECONDARY OUTCOMES:
Clinical worsening to critical COVID-19 illness | until Day 30
  Critical COVID-19 illness as a composite of admission to the intensive care unit (ICU), invasive ventilation, or death
Duration of supplemental oxygen therapy | until day 14
  Measured by duration of use of supplemental oxygen (if applicable)
Duration of mechanical ventilation (if applicable) | until day 30
  Measured by duration of use of mechanical ventilation
Duration of hospitalisation | until day 30
  Measured by duration of hospitalization
Proportion of participants with virologic clearance in nasopharyngeal swab RT-PCR | Day 14
  Presence or absence of SARS-CoV-2 Viral RNA in nasopharyngeal swab or lower respiratory secretions
C-reactive protein (CRP) level's reduction | Days 3, 5 and 8
  Reduction of C-reactive protein levels > 50% in comparison with PCR levels at the admission
Incidence of New Onset Lymphopenia | Through study completion, average of 15 days
  Incidence of new onset lymphopenia during hospitalization measured by blood draw
Direct bilirubin level's reduction | Measured in study Days 3, 5, and 8
  Reduction of mean direct bilirubin levels in comparison with levels at the admission
Side Effects | until day 14
  Differences in number of patients in study arms who experienced side effects

CONTACTS AND LOCATIONS:
Overall Officials: Dalva Poyares, PhD, Study Director — Associação Fundo de Incentivo a Pesquisa

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF